CLINICAL TRIAL: NCT03702140
Title: Examination How the Administration Period of Teriparatide Affects Bone Metabolism and Bone Mineral Density Prior to Denosumab Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shinshu University (Other)
Responsible Party: Principal Investigator, Yukio Nakamura, Lecturer at Shinshu University School of Medicine, Shinshu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PTH-DMAb 2018
Record Dates: First submitted 2018-10-08; First posted 2018-10-10 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Teriparatide

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TPTD 6M (Active Comparator)
  Interventions: Drug: "Teriparatide", "Forteo® or Teribon"
- TPTD 6-12M (Active Comparator)
  Interventions: Drug: "Teriparatide", "Forteo® or Teribon"
- TPTD 12-24M (Active Comparator)
  Interventions: Drug: "Teriparatide", "Forteo® or Teribon"

INTERVENTIONS:
Drug: "Teriparatide", "Forteo® or Teribon" — To examine the effects of terimaratide less than 6 months in osteoporosis

SUMMARY:
The aim of this study is to examine the efficacy and adverse events in the following 3 groups in osteoporosis patients:

1. The administration period of teriparatide is less than 6 months and thereafter, denosumab for 24 months.
2. The administration period of teriparatide is from 6 to 12 months and thereafter, denosumab for 24 months.
3. The administration period of teriparatide is more than 12 months and thereafter, denosumab for 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Osteoporotic patients who want to take teriparatide and denosumab

Exclusion Criteria:

* Patients who are allergic to teriparatide or denosumab Patients who are pregnant or breast-feedin

Ages: 20 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients are separately analyzed
Enrollment: 90 (Estimated)
Dates: Start 2018-10-09 (Actual); Primary Completion 2023-10-08 (Estimated); Study Completion 2025-10-08 (Estimated)

PRIMARY OUTCOMES:
Bone mineral density | Change from Baseline Values at 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Yukio Nakamura, Matsumoto, Nagano, Japan

IPD SHARING:
Plan to Share IPD: No